CLINICAL TRIAL: NCT04277494
Title: The Acute Effect of Cold Spray Application on the Mechanical Properties of the Quadriceps Muscle in Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-17/20
Record Dates: First submitted 2020-02-07; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-01

CONDITIONS: Cold; Spray; Muscle; Athletic Injuries
Keywords: cold; spray; muscle; Athletic Injuries
MeSH Terms: conditions — Common Cold; Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clorethyl cold spray® (Vapocoolant spray) (Experimental): 23 volunteer athletes who are studying at the Faculty of Health Sciences of Acıbadem University, between the ages of 18-23, with a subcutaneous fold thickness of the quadriceps muscle between 5 mm and 15 mm (Shadgan et al., 2015).
  From the anterior superior of the dominant legs to the spinal iliac, the upper part of the patella will be measured and the center point will be marked. Cold spray will be applied to this point and its surroundings. The ethyl chloride spray bottle will be kept approximately 30 cm from the skin. An ethyl chloride stream will be applied at a 45 ° angle for 15 seconds (Shadgan et al., 2015). Skin temperature and mechanical properties of muscle; will be measured before, immediately after, 2 minutes, 5 minutes and 15 minutes after cold application.
  Interventions: Other: Clorethyl cold spray® (Vapocoolant spray)

INTERVENTIONS:
Other: Clorethyl cold spray® (Vapocoolant spray) — From the anterior superior of the dominant legs to the spinal iliac, the upper part of the patella will be measured and the center point will be marked. Cold spray will be applied to this point and its surroundings. The ethyl chloride spray bottle will be kept approximately 30 cm from the skin. An ethyl chloride stream will be applied at a 45 ° angle for 15 seconds (Shadgan et al., 2015). Skin temperature and mechanical properties of muscle; will be measured before, immediately after, 2 minutes, 5 minutes and 15 minutes after cold application.

SUMMARY:
Vikocoolant spray, also known as cold spray; It is a form of cryotherapy (cold treatment) used in sports medicine, athletic training, sports competitions and rehabilitation environments. It has been demonstrated in the literature that local cold application may cause increased resistance to movement. It has been reported in some studies that muscle can change its mechanical properties in a short time. However, the effect of cold spray application on the mechanical properties of the muscle is unknown. Therefore, in the current study proposal, the investigators aim to investigate the acute effect of cold spray application on the mechanical properties of the quadriceps muscle in athletes.

DETAILED DESCRIPTION:
Tissue cooling (cryotherapy treatment) is a long-standing pain therapy for the treatment of acute injuries and during rehabilitation. It is used in addition to other treatments . The main purpose of cryotherapy is to cool the tissue temperature and is used in the clinic in the form of various cryotherapy modalities such as whole body cryotherapy, cold spray, cryotherapy clamps, frozen peas, cold water immersion, ice and cold packs . The first physiological response of cooling is a decrease in tissue temperature . Studies have shown that local cold application causes increased resistance to movement . Although it has been reported in animal studies conducted in vitro that muscle tissue shows high resistance to stretching after cooling down , only one study evaluating direct mechanical responses to muscles in human studies There. In this study carried out by Mustalampi et al., Parameter measurements indicating the mechanical properties of the muscle immediately after applying the cold pack applied locally to the quadriceps muscle for 20 minutes and after 15 minutes. As a result of the study, the muscle has become stiffer, less elastic in terms of mechanical properties and it has been shown that these changes do not completely recover after 15 minutes. It was also stated that careful warm-up should be recommended after cooling to normalize the mechanical properties of the muscle and prevent injury .

Also known as cold spray, vikocoolant spray is a form of cryotherapy used in sports medicine, athletic training and rehabilitation environments and is widely used in the world . Especially in field medicine, it is frequently used as the first treatment of sports injuries. However, as is often done, returning to the game and competition with the help of the emerging analgesia is inconvenient in terms of the treatment of injury . However, it is still used frequently due to ease of application. The use of cold spray as a therapeutic method is of particular interest, as it is typically applied for a much shorter time than other cryotherapy modes . It has been shown in the literature that local cold application can cause increased resistance to movement and it is reported that it can change the mechanical properties of the muscle in a short time. However, the effect of cold spray application on the mechanical properties of the muscle is unknown. Therefore, in the current study proposal, the investigators aim to investigate the acute effect of cold spray application on the mechanical properties of the quadriceps muscle in athletes.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer athletes between the ages of 18-25 with a subcutaneous fold thickness of the quadriceps muscle between 5 mm and 15 mm.
* Non-smoker
* No drug use

Exclusion Criteria:

Having any cardiovascular or peripheral vascular disease

* Known neuromuscular pathology history
* Having diabetes mellitus
* Having a history of lower limb pain and previous surgery
* A history of insensitivity to local heat or cold

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Estimated)
Dates: Start 2020-01-12 (Actual); Primary Completion 2020-02-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of skin temperature | Change from skin temperature at 0 minute, 2 minute, 15 minute post-spray
  For thermal imaging, a 120-9-90 pixel resolution FLIR E5 camera thermal camera (FLIR Systems AB, Sweden) will be used, and Color Palette iron will be selected to display images. The video will be taken from a distance of 1 m at a speed of 8 photos / s.
Evaluation of the mechanical properties of the muscle-1 | Change from mechanical properties at 0 minute, 2 minute, 15 minute post-spray
  Viscoelastic stiffness [N/m] will be measured in MyotonPro 3 (MYO, Tallin, Estonia).
Evaluation of the mechanical properties of the muscle-2 | Change from mechanical properties at 0 minute, 2 minute, 15 minute post-spray
  Oscillation frequency (Hz) will be measured in MyotonPro 3 (MYO, Tallin, Estonia).
Evaluation of the mechanical properties of the muscle-3 | Change from mechanical properties at 0 minute, 2 minute, 15 minute post-spray
  Mechanical stiffness (N/m)will be measured in MyotonPro 3 (MYO, Tallin, Estonia).

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mac Auley DC. Ice therapy: how good is the evidence? Int J Sports Med. 2001 Jul;22(5):379-84. doi: 10.1055/s-2001-15656. PMID 11510876
- [Background] Bizzini M, Mannion AF. Reliability of a new, hand-held device for assessing skeletal muscle stiffness. Clin Biomech (Bristol). 2003 Jun;18(5):459-61. doi: 10.1016/s0268-0033(03)00042-1. PMID 12763442
- [Background] Bleakley C, McDonough S, MacAuley D. The use of ice in the treatment of acute soft-tissue injury: a systematic review of randomized controlled trials. Am J Sports Med. 2004 Jan-Feb;32(1):251-61. doi: 10.1177/0363546503260757. PMID 14754753
- [Background] Enwemeka CS, Allen C, Avila P, Bina J, Konrade J, Munns S. Soft tissue thermodynamics before, during, and after cold pack therapy. Med Sci Sports Exerc. 2002 Jan;34(1):45-50. doi: 10.1097/00005768-200201000-00008. PMID 11782646
- [Background] Mustalampi S, Ylinen J, Kautiainen H, Weir A, Hakkinen A. Acute effects of cold pack on mechanical properties of the quadriceps muscle in healthy subjects. Phys Ther Sport. 2012 Nov;13(4):265-9. doi: 10.1016/j.ptsp.2012.02.001. Epub 2012 Apr 23. PMID 23068904